CLINICAL TRIAL: NCT02782897
Title: A Pilot Study of Safety and Efficacy of Intravenous Immunoglobulin Therapy in Patients With Acute Intracranial Hemorrhage
Brief Title: Intravenous Immunoglobulin for Acute Intracranial Hemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Wang (Other)
Responsible Party: Sponsor-Investigator, Wei Wang, Tongji Hospital, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016ncx01
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Intracranial Hemorrhage, Hypertensive
Keywords: intravenous immunoglobulin; intracerebral hemorrhage; perihematomal edema
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Cerebral Hemorrhage | interventions — Immunization, Passive; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIg group (Experimental): Participants will receive immunoglobulin therapy plus standard management. The first intravenous infusion of immunoglobulin must be given within 72 hours after the onset.
  Interventions: Drug: Immunoglobulin Therapy; Other: Standard management
- Control group (Other): Participants will receive standard management according to Chinese guidelines for intracerebral Hemorrhage.
  Interventions: Other: Standard management

INTERVENTIONS:
Drug: Immunoglobulin Therapy — Immunoglobulin is given intravenously 0.4 g/kg per day for five consecutive days.
  Other Names: Human Immunoglobulin (pH4) for Intravenous Injection
  Arms: IVIg group
Other: Standard management — Standard management includes: the use of mild sedation, blood pressure control, management of elevated intracranial pressure, glucose management, temperature management, airway maintenance, and management of medical complications.
  Other Names: Conventional treatment

SUMMARY:
This pilot study aims to investigate whether intravenous immunoglobulin is safe and effective in alleviating perihematomal edema and neurologic deficits in patients with intracranial hemorrhage.

DETAILED DESCRIPTION:
The trial consists of two groups: IVIg group and control group. Thirty patients will be recruited into IVIg group. Thirty Patients who are matched for age, gender, National Institutes of Health Stroke Scale scores, hematomal volumes, and locations of hematomas, will be selected into control group. Patients in control group just receive standard management, while those in IVIg group will receive standard management plus intravenous immunoglobulin therapy. The outcome assessor is blinded to the group assignments.

ELIGIBILITY:
Inclusion Criteria:

1. The first-ever primary supratentorial intracerebral basal ganglia hemorrhage 5-30ml.
2. 18-80 years old.
3. No longer than 72 hours from the acute ICH to medication.
4. Glasgow Coma Score ≥8.

Exclusion Criteria:

1. Occurrences of secondary intracerebral hemorrhage.
2. Significant past history of disability, modified Rankin Scale（mRS）≥1.
3. Currently taking antitumor drugs, immunosuppressive drugs, or immunomodulatory therapy.
4. Patients with pregnancy, Severe infection, severe heart dysfunction or renal and hepatic injuries.
5. Patients with contraindications for immunoglobulin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of the patients with mRS of 3 or more | 90 days after the onset of ICH

SECONDARY OUTCOMES:
Changes in hematoma volume | At baseline, 7 days, 14 days and 30 days after the onset
Change in peripheral edema volume | At baseline, 7 days, 14 days and 30 days after the onset
All-cause mortality | 90 days after the onset
mRS score | 30 days, 90 days after the onset
mBI score | 30 days, 90 days after the onset
Incidence of severe adverse events | 30 days, 90 days after the onset
Change in the levels of blood CRP, MMP-9, IL-6, TNF-alpha, and C3 | At baseline, 5 days after the first administration of immunoglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology, Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided